CLINICAL TRIAL: NCT05816200
Title: Comparative Analysis of Low-Level Light Therapy and Transcutaneous Electrical Nerve Stimulation for Burning Mouth: a Randomized Clinical Trial
Brief Title: Comparison Between Two Treatments for Burning Mouth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Cristianne Kalinne Santos Medeiros, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1274-3207; RBR-7fvcjkz (Registry Identifier: Brazilian Registration of Clinical Trials (ReBEC))
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Burning Mouth Syndrome
Keywords: Low-Level Light Therapy; Transcutaneous Electric Nerve Stimulation
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Low-Level Light Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Grupo TENS (Experimental): Participants with burning mouth underwent to transcutaneous electrical nerve stimulation
  Interventions: Device: Transcutaneous Electric Nerve Stimulation
- Grupo LLLT (Active Comparator): Participants with burning mouth underwent low-level laser therapy
  Interventions: Device: Low-Level Light Therapy

INTERVENTIONS:
Device: Low-Level Light Therapy — Punctual applications of infrared laser (L2) (power of 100mW, 808 nm, 6 joules of energy/60 seconds) in the affected region, keeping one centimeter of distance between the points, until the entire area of the complaint was irradiated. being held one session per week, totaling eight weeks of treatment at the end of the study.
  Other Names: Low Power Laser Therapy
  Arms: Grupo LLLT
Device: Transcutaneous Electric Nerve Stimulation — Using a device at a frequency of 50 Hertz with intensity modulated according to the patient's comfort ranging from 1 - 4 (pulse amplitude) with a duration of 25 minutes per session, with one session per week, totaling eight weeks of treatment at the end of the study. The device's self-adhesive electrodes were fixed on the participant's face, following the path of the trigeminal nerve branch on the side affected by pain and/or burning.
  Arms: Grupo TENS

SUMMARY:
Introduction: The management of patients with chronic burning mouth is a challenge in clinical dentistry. Objective: To compare the effect of Low Level Laser Therapy (LLLT) and Transcutaneous Electrical Nerve Stimulation (TENS) in the treatment of burning mouth. Materials and Methods: Randomized clinical trial consisting of 25 patients with burning mouth who were treated by TENS (n=12) and by LLLT (n=13). Treatment was carried out weekly for 8 weeks. Two-way ANOVA was used to verify whether there was a significant difference between times T0 (baseline), T1 (after the 4th treatment session), T2 (after the 8th treatment session) and T3 (30 days after the end of treatment) in in relation to symptoms, analyzed using the Visual Analog Scale, unstimulated salivary flow, xerostomia and dysgeusia with TENS and LLLT interventions.

DETAILED DESCRIPTION:
Experimental group: 20 participants with burning mouth were submitted to transcutaneous electrical nerve stimulation using a device at a frequency of 50 Hertz with intensity modulated according to the patient's comfort ranging from 1 - 4 (pulse amplitude) with a duration of 25 minutes per session, with one session per week, totaling eight weeks of treatment at the end of the study. The device's self-adhesive electrodes were fixed on the participant's face, following the path of the trigeminal nerve branch on the side affected by pain and/or burning.

Control group: 20 participants with burning mouth underwent low power laser therapy with punctual applications of infrared laser (L2) (power of 100mW, 808 nm, 6 joules of energy/60 seconds) in the affected region, keeping one centimeter of distance between the points, until the entire area of the complaint was irradiated. being held one session per week, totaling eight weeks of treatment at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or over
* Patients with burning sensation in the oral mucosa or recurrent dysesthetics daily for more than 2 hours a day for more than 3 months, without clinically evident causal lesions (IHS, 2018) were included in the study, as well as those who presented hyposalivation or some systemic alteration that could be related to a burning sensation in the oral mucosa

Exclusion Criteria:

• Patients who did not comply with the study treatment protocol.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Oliveira, PhD, Study Director — Universidade Federal do Rio Grande do Norte
Locations (1):
- Department of Dentistry, Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No
The article referring to this clinical trial is being edited for subsequent publication in a journal.

REFERENCES:
- [Result] Arduino PG, Cafaro A, Garrone M, Gambino A, Cabras M, Romagnoli E, Broccoletti R. A randomized pilot study to assess the safety and the value of low-level laser therapy versus clonazepam in patients with burning mouth syndrome. Lasers Med Sci. 2016 May;31(4):811-6. doi: 10.1007/s10103-016-1897-8. Epub 2016 Feb 12. PMID 26873501
- [Derived] Medeiros CKS, Serrao MDCPN, de Lima AAS, da Silveira EJD, de Oliveira PT. Comparative analysis of photobiomodulation therapy and transcutaneous electrical nerve stimulation for burning mouth: a randomized clinical trial. Clin Oral Investig. 2023 Oct;27(10):6157-6165. doi: 10.1007/s00784-023-05232-7. Epub 2023 Sep 1. PMID 37656286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of patients complaining of burning mouth treated at the Stomatology Service of the Department of Dentistry (DOD) at UFRN from April 2021 to February 2022.
Pre-assignment Details: Individuals who presented clinical changes in the oral mucosa such as erosive lichen planus, geographic tongue, infections, allergic reactions, trauma and injuries caused by physical or chemical agents were excluded.
Groups:
- Grupo LLLT: Participants with burning mouth underwent low-level laser therapy. One participant was excluded from this group for not completing the treatment protocol of the present study
  Low-Level Light Therapy: Punctual applications of infrared laser (L2) (power of 100mW, 808 nm, 6 joules of energy/60 seconds) in the affected region, keeping one centimeter of distance between the points, until the entire area of the complaint was irradiated. being held one session per week, totaling eight weeks of treatment at the end of the study.
Period: Overall Study
Arm/Group | Grupo TENS | Grupo LLLT
Started | 14 | 14
Completed | 12 | 13
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Grupo TENS | Grupo LLLT | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants] — The age of the participants was measured in years, from which the average age of the participants in each group was calculated.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 9 | 7 | 16
    >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.36 (10.56) | 61.36 (10.40) | 59.86 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was measured based on the Brazilian Institute of Geography and Statistics (IBGE) classification for the ethnic or racial denomination of people in Brazil. This classification includes the terms: black, brown, yellow, indigenous or white.
  Participants
    Baseline (T0): White | 10 | 07 | 17
    Baseline (T0): Brown | 2 | 6 | 8
Region of Enrollment [Count of Participants; unit: Participants] — This randomized clinical trial involved patients with burning mouth seen at the Stomatology Service of the Department of Dentistry, Federal University of Rio Grande do Norte (UFRN), Natal, RN, Brazil. Population: Patients older than 18 years who had a burning or dysesthetic sensation in the oral mucosa that recurred daily for more than 2 h per day for more than 3 months, in the absence of clinically evident causal lesions, were included in the study. We also included patients with hyposalivation or any systemic alteration that could be related to a burning sensation in the oral mucosa.
  Participants
    Brazil | 12 | 13 | 25
Painful symptoms [Mean (Standard Deviation); unit: units on a scale] — Pain/burning was the primary outcome and was measured on a visual analogue scale (VAS; 0-10 cm). Patients were asked to choose a number from 0 to 10 on the scale to describe the level of intensity of their symptoms, with higher values representing a worse outcome.
  units on a scale | 7.58 (2.64) | 6.92 (2.54) | 7.39 (2.48)

OUTCOME MEASURES:

1. Primary Outcome: Painful Symptoms
Description: Changes in the intensity of pain/burning was determined by Visual Analogue Scale. Possible scores range from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline (T0), after the 4th treatment session (4 weeks), after the 8th treatment session (8 weeks). ), 30 days after the end of treatment (8 weeks + 30 days).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Grupo TENS | Grupo LLLT
Number analyzed (Participants) | 12 | 13
score on a scale
  T0 | 7.58 (2.64) | 6.92 (2.54)
  T1 | 5.08 (2.94) | 5.33 (3.23)
  T2 | 3.17 (2.48) | 4.50 (2.88)
  T3 | 5.75 (2.49) | 3.75 (3.08)

2. Secondary Outcome: Salivary Flow
Description: The unstimulated salivary flow rate will be determined by the ratio volume of saliva collected, expressed in millimeters per minute (ml/min).
Time Frame: Baseline (T0), after the 4th treatment session (4 weeks), after the 8th treatment session (8 weeks). ), 30 days after the end of treatment (8 weeks + 30 days
Measure: Mean (Standard Deviation); unit: average of ml collected per minute
Arm/Group | Grupo TENS | Grupo LLLT
Number analyzed (Participants) | 12 | 13
average of ml collected per minute
  T0 | 0.32 (0.23) | 0.27 (0.20)
  T1 | 0.22 (0.08) | 0.30 (0.30)
  T2 | 0.36 (0.22) | 0.22 (0.13)
  T3 | 0.30 (0.36) | 0.24 (0.14)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Grupo LLLT: Participants with burning mouth underwent low-level laser therapy. Low-Level Light Therapy: Punctual applications of infrared laser (L2) (power of 100mW, 808 nm, 6 joules of energy/60 seconds) in the affected region, keeping one centimeter of distance between the points, until the entire area of the complaint was irradiated. being held one session per week, totaling eight weeks of treatment at the end of the study.
Arm/Group | Grupo LLLT | Grupo TENS
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT05816200/Prot_SAP_001.pdf